CLINICAL TRIAL: NCT07104253
Title: Establishing Feasibility of Transbronchial Cryoablation With an In-Development Cryoprobe: An Ex-Vivo Human Lung Model
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Endocision Technologies Inc. (Industry)
Collaborators: Centre de Recherche du Centre Hospitalier de l'Université de Montréal (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2025-12805
Record Dates: First submitted 2025-07-11; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Lung Cancer
Keywords: Lung Cancer; Transbronchial Ablation; Cryoablation
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ex Vivo Cryo (Experimental): Multiple procedures will be performed to each model in order to accomplish the objectives of the study. Tissue samples will be taken from the models and images will be performed. This will allow us to determine which configuration is the optimal for obtaining the more effective and stable models that could offer the best quality specimens as well.
  Interventions: Device: Ex vivo cryo-ablation

INTERVENTIONS:
Device: Ex vivo cryo-ablation — With informed consent obtained prior to transplantation, explanted lungs from patients undergoing lung transplantation will be obtained. The organs will be placed in an acrylic box and will be perfused at a temperature of 37 Celsius degrees. The lungs will be mechanically ventilated connected by an endotracheal tube size 7 inserted in the bronchus with the balloon inflated and a silk suture providing a hermetic closure proximal to the balloon. The cryocatheter will be inserted in the lungs and cryoablation will be performed with varying freeze-thaw cycles to confirm design and operating specifications of the device.

SUMMARY:
Demonstrate the application of in-development cryogenic catheters for the ablation of pulmonary lesions.

DETAILED DESCRIPTION:
Surgical resection is the current gold standard for curative treatment of pulmonary lesions. For patients ineligible for surgical resection, transthoracic percutaneous ablation is sometimes used. Albeit the use of minimally techniques for both surgery and ablation, these interventions are associated with a high risk of complication. To reduce associated risks, transbronchial interventions have been proposed as promising alternatives. However, currently available transbronchial ablation technologies may present significant risks of bleeding or lack clinical evidence with regards to efficacy. When considering potential alternatives, promising results have been achieved using cryotechnology for cryoablation. However, the feasibility of a transbronchial cryoablation device and its thermal performance at varying freeze-thaw cycles in a clinical setting is unknown. The investigators aim to demonstrate the application of in-development transbronchial cryogenic catheters for the ablation of pulmonary lesions.

The investigators aim to confirm the design and operating specifications of an in-development cryogenic catheters for the ablation of pulmonary lesions and investigate the thermal performance of the catheter.

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing lung transplant surgery

Exclusion Criteria:

Organ donors eligible to donate lungs for transplantation Healthy individuals Patients with ongoing pulmonary infection at the time of transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Tissue temperature at 5 mm from the probe over intervention time | 48 months
  Measuring the temperature is and indicator of thermal cooling power and is required to confirm the design and operating specifications of the cryocatheter.
Tissue temperature at 10 mm from the probe over intervention time | 48 months
  Measuring the temperature is and indicator of thermal cooling power and is required to confirm the design and operating specifications of the cryocatheter.
Tissue temperature at 15 mm from the probe over intervention time | 48 Months
  Measuring the temperature is and indicator of thermal cooling power and is required to confirm the design and operating specifications of the cryocatheter.

SECONDARY OUTCOMES:
Iceball size | 48 months
  Measurement of the major axis in mm of the resulting iceball to confirm the design and operating specifications of the cryocatheter

IPD SHARING:
Plan to Share IPD: No